CLINICAL TRIAL: NCT05047991
Title: A Multicenter, Randomized, Open-lable, Parallel-controlled, Phase II Study to Evaluate the Differences of Safety and Efficacy of Irinotecan Liposome Injection-containing Regimens Versus Nab-paclitaxel Plus Gemcitabine in Patients With Previously Untreated, Metastatic Pancreatic Adenocarcinoma
Brief Title: Study of Irinotecan Liposome Injection-containing Regimens Versus Nab-paclitaxel Plus Gemcitabine in Patients With Previously Untreated, Metastatic Pancreatic Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE072-CSP-004
Record Dates: First submitted 2021-08-26; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Pancreatic Cancer Non-resectable; Pancreatic Cancer Metastatic
MeSH Terms: interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin; Oxaliplatin; Taxes; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Irinotecan Liposome Injection + 5-FU/LV + Oxaliplatin (Experimental): The patients in cohort 1 will receive irinotecan liposome injection combined with 5-fluorouracil (5-FU), leucovorin(LV) and oxaliplatin intravenously on day 1 and day 15 of every 28-day cycle until disease progression or unacceptable toxicity, or termination of the study due to other reasons.
  Interventions: Drug: Irinotecan Liposome Injection; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- Cohort 2: Nab-paclitaxel + Gemcitabine (Active Comparator): The patients in cohort 2 will receive nab-paclitaxel and gemcitabine intravenously on day 1、day 8 and day 15 of every 28-day cycle until disease progression or unacceptable toxicity, or termination of the study due to other reasons.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Irinotecan Liposome Injection — Irinotecan Liposome Injection, intravenously, over 90 min on day 1and day 15 of every 28-day cycle
  Arms: Cohort 1: Irinotecan Liposome Injection + 5-FU/LV + Oxaliplatin
Drug: Fluorouracil — 5-Fluorouracil (5-Fu), intravenously, over 46 h on day 1 and day 15 of every 28-day cycle
  Arms: Cohort 1: Irinotecan Liposome Injection + 5-FU/LV + Oxaliplatin
Drug: Leucovorin — Leucovorin (LV), intravenously, over 30 min on day 1 and day 15 of every 28-day cycle
  Arms: Cohort 1: Irinotecan Liposome Injection + 5-FU/LV + Oxaliplatin
Drug: Oxaliplatin — Oxaliplatin, intravenously, over 2 h on day 1 and day 15 of every 28-day cycle
  Arms: Cohort 1: Irinotecan Liposome Injection + 5-FU/LV + Oxaliplatin
Drug: Nab paclitaxel — Paclitaxel (albumin bound), intravenously, over 30 min on day 1, day 8 and day 15 of every 28-day cycle
  Arms: Cohort 2: Nab-paclitaxel + Gemcitabine
Drug: Gemcitabine — Gemcitabine, intravenously, over 30 min on day 1, day 8 and day 15 of every 28-day cycle
  Arms: Cohort 2: Nab-paclitaxel + Gemcitabine

SUMMARY:
This is a multicenter, randomized, open-lable, parallel-controlled phase II study of irinotecan liposome injection-containing regimens versus nab-paclitaxel plus gemcitabine in patients with previously untreated, metastatic pancreatic adenocarcinoma. The purpose of this study is to evaluate the differences of safety and efficacy of irinotecan liposome injection-containing regimens versus nab-paclitaxel plus gemcitabine in patients with previously untreated, metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
This is a multicentre randomized, open-label, parallel-controlled, phase II study to evaluate the efficacy and safety of irinotecan liposome injection-containing regimens. Eligible patients will be randomly divided into two cohorts at a ratio of 2:1. The patients in cohort 1 (the experimental group) will receive irinotecan liposome injection combined with 5-fluorouracil (5-FU), leucovorin (LV) and oxaliplatin.The patients in cohort 2 (the control group) will receive nab-paclitaxel plus gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years old (inclusive), regardless of gender;
2. Histologically or cytologically confirmed unresectable, locally advanced, or metastatic pancreatic adenocarcinoma;
3. At least one measurable lesion according to RECIST 1.1.
4. No prior systemic anti-tumor therapy, except those with disease progression more than 6 months after adjuvant therapy or neoadjuvant therapy;
5. Patients with prior local treatment (radical radiotherapy or radical chemoradiotherapy, etc.) may be enrolled provided that the local treatment does not involve the target lesion, or the target lesion is within the treatment area, but the size has increased more than 20% since the post-treatment evaluation, and also must be completed at least 4 weeks before the first administration of the study drug, palliative decompensated radiotherapy (such as bone metastases) must be completed at least 2 weeks before the first administration of the study drug;
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1;
7. Life expectancy >3 months;
8. Adverse reactions must recover to grade 1 or baseline according to CTCAE 5.0 (except for toxicity such as alopecia, grade 2 or less sensory neuropathy, etc., which have been judged no safety risk by investigators).
9. Patients should not receive cell growth factors or blood and platelet transfusion within 7 days before the initiate administration of study drug, and laboratory test must meet the following criteria:

   neutrophile count ≥1.5×10^9/L; platelet count ≥100×10^9/L; hemoglobin ≥90 g/L or ≥5.6 mmol/L; serum creatinine ≤1×ULN or creatinine clearance rate must be ≥ 50 mL/min when serum creatinine >1.0×ULN; total bilirubin ≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN or ≤5×ULN if intrahepatic lesions exist; Albumin ≥3 g/dL.
10. Activated Partial Thromboplastin Time (APTT), International Normalized Ratio (INR) and prothrombin time (PT) ≤1.5 × ULN for patients not receiving therapeutic anticoagulation.
11. According to the related guidelines, patients with HBV DNA or HBsAg and/or anti-HBC positive must receive prophylactic treatment (at least one week before the initial administration of the study drug) and take antiviral drugs in stable dose (e.g., entecavir, tenofovir, or lamivudine; No adefovir or interferon are allowed) at study entry with planned monitoring and management, including baseline HBV DNA levels. Patient receiving active hepatitis C virus (HCV) treatment must use astable dose of drugs at study entry and be subject to planned monitoring and management according to antiviral drug guidelines;
12. Female patients with reproductive potential must agree to use adequate contraception from the signing of informed consent to at least 6 months after the study completion and have a negative serum pregnancy test within 3 days before enrollment, and must be non-lactating. Male patients must agree to use medically approved contraception during the study period and for 6 months after the study completion;
13. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Patients with acinar cell carcinoma, pancreatoblastoma, solid pseudopapillary tumor and pancreatic neuroendocrine tumor;
2. Patients with definitive diagnosis of CNS metastasis;
3. Patients with hepatic encephalopathy at screening;
4. Patients with clinically symptomatic ascites requiring puncture or drainage or who have received ascites drainage within the past 3 months, except for those with only a small amount of ascites on imaging but no clinical symptoms;
5. Uncontrolled third lacunar effusion other than ascites (e.g., large pleural or pericardial effusion) within 4 weeks before the first administration of the test drug;
6. Previous malignancies in the past five years (except radically resected and non-recurring basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder carcinoma, local prostate carcinoma, carcinoma in situ of cervical, or other carcinoma in situ);
7. Patients with partial or complete biliary obstruction who has not relieved by active treatment;
8. History of serious cardiovascular disease, including but not limited to:

1) Acute myocardial infarction, unstable angina pectoris, coronary angioplasty, stroke, severe pulmonary embolism; 2) New York Heart Association class grade III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50%; 3) Poorly controlled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure≥ 95 mmHg) with optimal treatment; 4) Ventricular arrhythmia; 5) Patients with prolonged QT/QTc interval in baseline electrocardiogram (ECG) (QTcF > 480 ms, Fridericia formula: QTcF = QT/(RR^0.33), RR = 60/heart rate); 6) Patients with clinically significant abnormal electrocardiogram (ECG) according to the investigator's assessment.

9.Patients with uncontrolled active bleeding.

10.Patients with known interstitial lung disease;

11.Patients with known peripheral neuropathy (CTCAE grade 3 or 4);

12.Patients with severe lung, liver, kidney, endocrine, immune system, skin or musculoskeletal diseases within 3 months prior to the first dose and who are not suitable for enrollment in the opinion of the investigator;

13.Patients who are at risk of active infection or have active infection that may affect the results of the study (such as severe pneumonia requiring hospitalization, bacteremia, acute bacterial infection, infectious complications, tuberculosis, active HIV infection, etc.) or who, in the judgment of the investigator, are not suitable for participation in this clinical trial. Active hepatitis B virus is defined as HBV DNA≥10^4 copies or ≥ 2000 IU/mL; active hepatitis C virus or active HIV infection is defined as HCV-RNA positive;

14.Gastrointestinal diseases of clinical significance, such as bleeding, inflammation, obstruction, >grade 1 diarrhea, malabsorption syndrome, diseases significantly affecting gastrointestinal function, gastric or small bowel resection, etc;

15.Patients with known to have dihydropyrimidine dehydrogenase (low activity) or deficiency;

16.Patients with definite Gilbert syndrome;

17.History of explicit neurological or psychiatric disorders, including epilepsy or dementia;

18.Patients with known alcohol or drug dependence.

19.Patients who have concomitant use of strong CYP3A4 inducers within 2 weeks prior to the first dose, or strong CYP3A4 inhibitors or strong UGT1A1 inhibitors within 1 week prior to the first dose;

20.Patients who have required systemic glucocorticoids (prednisone >10 mg/day or equivalent dose of the similar drugs) or other immunosuppressive agents within 14 days before the first dose of the study drug. Except for treatment with local, ocular, intra-articular, intranasal, and inhaled glucocorticoids in the absence of active autoimmune disease, short-term preventive treatment with glucocorticoids (e.g., prevention of contrast allergy);

21.Patients who have major organ surgery (except for needle biopsy, central venous catheterization, port-cath, stenting to relieve biliary obstruction, and percutaneous hepatic biliary drainage, cholecystostomy) or selective operation plan were performed within 4 weeks before the first dose of the study drug;

22.Patients with known allergy to irinotecan liposome injection, other liposome products, oxaliplatin, 5-fluorouracil, leucovorin, Nab-paclitaxel, other albumin products, gemcitabine or any of the ingredients in the above products.;

23. Patients who are not suitable for this study as determined by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to twelve months after the last patient's first administration
  Time from date of the first dose to date of recorded disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to twelve months after the last patient's first administration
  The percentage of patients who achieve a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
Overall survival (OS) | Up to twelve months after the last patient's first administration
  Time from date of the first dose to date of death from any cause.
Disease Control Rate (DCR) | Up to twelve months after the last patient's first administration
  The percentage of patients who achieve a CR, PR or stable disease (SD) based on the RECIST 1.1.
Duration of Response (DOR) | Up to twelve months after the last patient's first administration
  Time from first documented response (CR or PR whichever occurs first, based on investigator's assessment per RECIST 1.1) to date of disease progression or death due to any cause, whichever occurs first.
Incidence of treatment-related adverse events (AEs) and serious adverse events (SAEs) | Up to twelve months after the last patient's first administration
  The AEs and SAEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0.
Peak Plasma Concentration | Day 0 to Day 7 of circle 1
  Cmax
Area under the plasma concentration versus time curve | Day 0 to Day 7 of circle 1
  AUC
UGT1A1 | Within 3 days before the first dose
  UGT1A1 gene polymorphism

IPD SHARING:
Plan to Share IPD: No